CLINICAL TRIAL: NCT05105945
Title: A Randomized, Controlled, Multi-center Clinical Study on the Efficacy of Single-port Inflatable Mediastinoscopy Combined With Laparoscopic-assisted Small Incision Surgery and Thoracoscopy Combined With Laparoscopic Surgery for Radical Esophagectomy
Brief Title: Clinical Study on the Efficacy of Single-port Inflatable Mediastinoscopy Combined With Laparoscopic-assisted Small Incision Surgery and Thoracoscopy Combined With Laparoscopic Surgery for Radical Esophagectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: General Hospital of Ningxia Medical University (Other); Beijing Chao Yang Hospital (Other); West China Hospital (Other); Shanghai Chest Hospital (Other); Peking University Cancer Hospital & Institute (Other); The First Affiliated Hospital of Nanchang University (Other); Changzhi Medical College (Other); Zhangzhou Affiliated Hospital of Fujian Medical University (Other); Harbin Medical University (Other); Hubei Cancer Hospital (Other); Jining First People's Hospital (Other); Jiangsu Cancer Institute & Hospital (Other); Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZDWY.XXW.005
Record Dates: First submitted 2021-09-16; First posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-08

CONDITIONS: Esophageal Cancer
Keywords: Minimally invasive surgery
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Laparoscopy

STUDY DESIGN:
Intervention Model Description: The Logrank method was used to compare the difference in survival time between the two groups of patients. According to previous literature data, it is estimated that the DFS of the control group is 18 months. Assuming that the DFS of the test group can be extended to 21.6 months (corresponding HR=1.20), the test requires 1048 patients (524 in each group) to achieve α=0.05 This difference can be detected with 80% confidence at the (two-sided) significance level. The trial plans to enroll for 48 months, follow up for 60 months, and conduct a final analysis when 944 patients have tumor progression (recurrence or metastasis). It is estimated that the drop-off rate of patients in the experimental group and the control group is 10%, so 1164 (524×2÷0.9=1164) patients need to be enrolled in the final group.
  Significance Level：0.05
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single port inflatable mediastinoscope and synchronized laparoscopic radical resection (Experimental): Detailed surgical procedures and related instructions have been published in "Single-Port Inflatable Mediastinoscopy Combined With Laparoscopic-Assisted Small Incision Surgery for Radical Esophagectomy Is an Effective and Safe Treatment for Esophageal Cancer" J Gastrointest Surg. 2019 Aug;23(8):1533-1540. doi: 10.1007/s11605-018-04069-w. Epub 2019 Jan 11.
  Interventions: Procedure: Single-Port Inflatable Mediastinoscopy Combined With Laparoscopic-Assisted Small Incision Surgery
- Thoracoscopy combined with laparoscopic radical resection (Active Comparator): Patients will receive a standardized thoracoscopy and laparoscopy combined radical esophageal cancer surgery
  Interventions: Procedure: Thoracoscopy Combined With Laparoscopic Surgery

INTERVENTIONS:
Procedure: Single-Port Inflatable Mediastinoscopy Combined With Laparoscopic-Assisted Small Incision Surgery — Single-Port Inflatable Mediastinoscopy Combined With Laparoscopic-Assisted Small Incision Surgery dissects, dissociates and removes the esophagus in the mediastinum through an inflatable endoscopy. Detailed surgical procedures and related instructions have been published in "Single-Port Inflatable Mediastinoscopy Combined With Laparoscopic-Assisted Small Incision Surgery for Radical Esophagectomy Is an Effective and Safe Treatment for Esophageal Cancer" J Gastrointest Surg. 2019 Aug;23(8):1533-1540. doi: 10.1007/s11605-018-04069-w. Epub 2019 Jan 11.
  Arms: Single port inflatable mediastinoscope and synchronized laparoscopic radical resection
Procedure: Thoracoscopy Combined With Laparoscopic Surgery — Patients will receive a standardized thoracoscopy and laparoscopy combined radical esophageal cancer surgery
  Arms: Thoracoscopy combined with laparoscopic radical resection

SUMMARY:
We previously developed a novel non-trans thoracic esophagectomy, the single-port inflatable mediastinoscopy combined with laparoscopy for the radical esophagectomy of esophageal cancer.This study is evaluating the feasibility and safety of radical resection of single-port inflatable mediastinal mirror synchronization with laparoscopic esophageal carcinoma, as well as the clinical value of the radical resection of single-port inflatable mediastinal mirror synchronization with laparoscopic esophageal carcinoma as a new minimally invasive operation for esophageal carcinoma.

DETAILED DESCRIPTION:
To reduce postoperative pulmonary complications, considerable efforts have been made to develop the nontransthoracic esophagectomy for esophageal cancer. For instance, esophageal stripping and transhiatal esophagectomy are the nontransthoracic operations developed for treatment for esophageal cancer. These methods possess several advantages, including non-thoracotomy, less postoperative pain, less postoperative cardiac and pulmonary complications, and safer for elderly patients. However, these two methods are limited with the poor surgical view, poor mediastinal lymph node dissection (especially upper mediastinal lymph nodes), and high risk of bleeding.

In 2015 and 2016, Prof. Fujiwara has developed novel surgical methods on the dissection of upper mediastinal lymph nodes using single-port mediastinoscopy through the cervical incision and the lower mediastinal lymph nodes (including the subcarinal lymph nodes) by laparoscopy, respectively.For the first time, non-transthoracic radical resection of esophageal cancer could be achieved along with the dissection of all the mediastinal lymph nodes. Based on the Fujiwara's method, we further improved this surgical method to the"single-port inflatable mediastinoscopy combined with laparoscopy for the radical treatment of esophageal cancer"and has successfully performed this novel surgical method for the first case in March 2016. We have completed over 200 cases of radical resection of esophageal carcinoma using this novel surgical technique from May 2016 to August 2021.

This is a prospective, multicenter, open clinical study in which 1164 patients (including 10% drop-off rate) who require surgical treatment are scheduled to be included in the study. Prior to any screening process, each subject / legal guardian should sign the informed consent form. Screening tests are used to determine whether each subject is eligible for the study. Eligible subjects who meet the standard will be treated with radical resection of single-hole inflatable mediastinal mirror synchronization with laparoscopic esophageal carcinoma and followed up until 5 years postoperatively. Primary study outcome are the prioperative complication rate and the number of intraoperative lymph node dissection.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old ≤ age ≤ 75 years old, no gender limit;
2. Patients who are diagnosed as esophageal malignant tumor by cytology or histology, and agree to undergo surgical treatment;
3. The preoperative clinical tumor staging is T1-2N0-1M0 patients; or T3N1-2M0 patients undergo neoadjuvant treatment (neoadjuvant chemotherapy, neoadjuvant chemoradiation, neoadjuvant radiotherapy, neoadjuvant chemotherapy and immunotherapy, neoadjuvant radiotherapy and immunotherapy After treatment), assess the tumor to achieve partial response (PR) and surgical resection is feasible;
4. The tumor is located in the thoracic esophagus;
5. The tumor has not invaded the surrounding vital organs and has metastasized far away;
6. The function of major organs is basically normal: general anesthesia is acceptable for lung function; NYHA grade of heart function is 0~1;
7. Voluntarily sign an informed consent form before the study. The patient and/or his legal representative have the ability to fully understand the content, process and possible adverse reactions of the experiment, and enable the patient to comply with the visits stipulated in the plan;

Exclusion Criteria:

1. People who suffer from other malignant tumors at the same time;
2. Patients with a history of esophagus or gastrectomy;
3. Patients with a history of mediastinal surgery or extensive abdominal cavity adhesion;
4. Patients with basic diseases such as cardiovascular and cerebrovascular diseases;
5. People suffering from mental, mental or neurological diseases;
6. Patients with cachexia and severe malnutrition who cannot tolerate surgery;
7. Recent recurrence of gastric ulcer, history of gastric bleeding and other serious underlying diseases;
8. Patients with surgical contraindications such as blood coagulation dysfunction, HIV antibody positive, and poorly controlled clinically severe infections;
9. Patients with other comorbid diseases (such as liver and kidney function abnormalities, etc.) or concomitant medications, which may have an impact on the results of this study based on the judgment of the investigator.
10. Patients who have participated in other clinical studies;
11. Others judged by the investigator to be unsuitable to participate in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1164 (Estimated)
Dates: Start 2021-11-11 (Estimated); Primary Completion 2027-12-28 (Estimated); Study Completion 2028-12-28 (Estimated)

PRIMARY OUTCOMES:
Perioperative incidence of cardiopulmonary complications | Through operation completion, an average of 12 days
  Perioperative complications include: pulmonary infection, respiratory failure, managed pleural effusion, heart failure, myocardial infarction, managed arrhythmia, anastomotic fistula or gastric fistula, recurrent laryngeal nerve injury, chylothorax, unscheduled reoperation
disease-free survival（DFS） | After surgery-related treatment until the tumor recurrence，assessed up to 5 years
  The period after Operation treatment [tumor eliminated] when no disease can be detected
overall survival（OS） | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years
  When the precise cause of Esophageal cancer death is not specified, this is called the overall survival rate or observed survival rate. Doctors use mean overall survival rates to estimate the patient's prognosis. This is often expressed over standard time periods, like one, five, and ten years.

SECONDARY OUTCOMES:
intraoperative blood loss | During the operation, an average of 2 hours
  Calculation of intraoperative bleeding with ml/kg
Operation time | During the operation, an average of 2 hours
  Calculate the operating time in minutes
Proportion of patients who converted to thoracotomy and laparotomy | During the operation, an average of 2 hours
  The ratio of the number of patients converted to thoracotomy or laparotomy to the total number of patients undergoing surgery
Intraoperative mortality rate | During the operation, an average of 2 hours
  The ratio of the number of patients who died during the operation to the number of patients who underwent the operation
Postoperative hospital stay | Through postoperative hospital stay, an average of 4 days
  The days of postoperative hospitalization
Postoperative pain score | An average of 3 days after the operation
  Daily pain scores were recorded by VAS (Visual Analogue Scale/Score) 1-3 days after operation
Postoperative admission time to ICU | An average of 3 days after the operation
  If the patient needs to be transferred to ICU after operation, stay in icu monitoring time should be observed
Postoperative drainage | An average of 3 days after the operation
  Total postoperative thoracic or mediastinal drainage (ml/kg)
Postoperative retention time of various types of drainage tubes | An average of 3 days after the operation
  The retention time of different types of drainage tube
Number of lymph nodes removed during surgery | Pathology report time, an average of 4 days
  The number of dissected lymph nodes reported in the postoperative pathology report

CONTACTS AND LOCATIONS:
Overall Officials: Liu Shaoxuan, Study Chair — Office of clinical research center
Locations (1):
- The Fifth Affiliated Hospital of Sun Yat-sen University, Zhuhai, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Choi AR, Chon NR, Youn YH, Paik HC, Kim YH, Park H. Esophageal cancer in esophageal diverticula associated with achalasia. Clin Endosc. 2015 Jan;48(1):70-3. doi: 10.5946/ce.2015.48.1.70. Epub 2015 Jan 31. PMID 25674530
- [Result] Luketich JD, Pennathur A, Franchetti Y, Catalano PJ, Swanson S, Sugarbaker DJ, De Hoyos A, Maddaus MA, Nguyen NT, Benson AB, Fernando HC. Minimally invasive esophagectomy: results of a prospective phase II multicenter trial-the eastern cooperative oncology group (E2202) study. Ann Surg. 2015 Apr;261(4):702-7. doi: 10.1097/SLA.0000000000000993. PMID 25575253
- [Result] Wang X, Li X, Cheng H, Zhang B, Zhong H, Wang R, Zhong B, Cao Q. Single-Port Inflatable Mediastinoscopy Combined With Laparoscopic-Assisted Small Incision Surgery for Radical Esophagectomy Is an Effective and Safe Treatment for Esophageal Cancer. J Gastrointest Surg. 2019 Aug;23(8):1533-1540. doi: 10.1007/s11605-018-04069-w. Epub 2019 Jan 11. PMID 30635830
- [Result] Fujiwara H, Shiozaki A, Konishi H, Kosuga T, Komatsu S, Ichikawa D, Okamoto K, Otsuji E. Single-Port Mediastinoscopic Lymphadenectomy Along the Left Recurrent Laryngeal Nerve. Ann Thorac Surg. 2015 Sep;100(3):1115-7. doi: 10.1016/j.athoracsur.2015.03.122. PMID 26354650
- [Result] Fujiwara H, Shiozaki A, Konishi H, Komatsu S, Kubota T, Ichikawa D, Okamoto K, Morimura R, Murayama Y, Kuriu Y, Ikoma H, Nakanishi M, Sakakura C, Otsuji E. Hand-assisted laparoscopic transhiatal esophagectomy with a systematic procedure for en bloc infracarinal lymph node dissection. Dis Esophagus. 2016 Feb-Mar;29(2):131-8. doi: 10.1111/dote.12303. Epub 2014 Dec 9. PMID 25487303